CLINICAL TRIAL: NCT05458921
Title: Study CARPUS : " Development of Automated Real-time Algorithms for Detection of Dislocation of the Carpus "
Brief Title: Development of Automated Real-time Algorithms for Detection of Dislocation of the Carpus
Acronym: CARPUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8559
Record Dates: First submitted 2022-07-08; First posted 2022-07-14 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Perilunate Dislocation
Keywords: Perilunate dislocation; Carpus dislocation; Radiocarpal osteoarthritis; mid-carpal osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Perilunate dislocation of the carpus is a serious lesion of the wrist which is defined by a total loss of contact of the articular surfaces capito-lunar, scapholunate and lunate-triquetral. Rare by its frequency, it represents 5 to 10% of traumatic injuries of the wrist.

Perilunate wrist dislocation is a rare injury that goes unnoticed in 25% of cases. Even with surgical treatment, 50-100% of patients will develop radiocarpal and/or midcarpal osteoarthritis.

ELIGIBILITY:
Inclusion criteria :

* Major subjects (≥18 years old)
* Treated at the University Hospitals of Strasbourg for a carpal dislocation
* Presence of carpal radiographs that may indicate the presence of a lesion
* Subjects who have not expressed their opposition, after information, to the re-use of their data for the purposes of this research

Exclusion criteria :

* Subject having expressed his opposition to participate in the study
* Subject under legal protection, guardianship or curatorship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subjects (≥18 years old) treated at the University Hospitals of Strasbourg for a carpal dislocation between 01/01/2012 and 31/12/2022.
Sampling Method: Non-Probability Sample
Enrollment: 10100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of carpal X-rays for the development of an algorithm to automatically identify the presence of pathology in the carpal anatomical area | Files analysed retrospectively from January 01, 2012 to December 31, 2022 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Philippe LIVERNEAUX, MD, PhD, Principal Investigator — Service de Chirurgie de la main - CHU de Strasbourg - France
Locations (1):
- Service de Chirurgie de la main - CHU de Strasbourg - France, Strasbourg, France